CLINICAL TRIAL: NCT04389489
Title: Evaluation of Pregnant Women Diagnosed With COVID-19 Using Carol Postpartum Sexual Function and Dyspareunia Scale
Brief Title: Postpartum Sexual Function in Pregnant Women With COVID-19
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Aldikactioglu Talmac, MD, Specialist of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: MTalmacCarol
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Dyspareunia; Postpartum Period
Keywords: Postpartum Period; Dyspareunia; COVID-19
MeSH Terms: conditions — COVID-19; Dyspareunia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19: Pregnant women with COVID-19 who have given birth
- Control: Healthy pregnant women who have given birth

SUMMARY:
The aim of this study is to identify women with postpartum sexual dysfunction and dyspareunia risk in the early period and to use the treatment and care services they need effectively. Our secondary aim is to reveal the difference in sexual life in the postpartum period between healthy pregnant women and pregnant women diagnosed with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Patient with COVID-19

Exclusion Criteria:

* Those with known sexual dysfunction disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In the reproductive age between 18-45 years old, two groups of 70 people will be selected, consisting of puerperant diagnosed with COVID-19 and healthy puerperant. Patients who have cesarean or vaginal delivery at the end of the study group, who do not have sexual intercourse dysfunction for another reason (such as Stage 3-4 perineal injury, vaginismus) will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of pregnant women diagnosed with COVID-19 using Carol Postpartum Sexual Function and Dyspareunia Scale | 3 months
  In the study planned to be carried out, it is aimed to identify women at risk of postpartum sexual dysfunction and dyspareunia early and benefit from the treatment and care services they need effectively.

SECONDARY OUTCOMES:
Evaluation of pregnant women diagnosed with COVID-19 using Carol Postpartum Sexual Function and Dyspareunia Scale | 3 Months
  To reveal the difference in sexual life in postpartum period between healthy pregnant women and pregnant women diagnosed with COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Halkali, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez-Lapeyrere C, Serna-Gomez N, Hernandez-Lopez AB, Perez-Garcia MF, Tejeda-Esteban A, Solis-Munoz M. The development and validation of a new postpartum sexual function and dyspareunia assessment tool: The Carol Scale. Midwifery. 2018 Mar;58:27-36. doi: 10.1016/j.midw.2017.11.008. Epub 2017 Dec 6. PMID 29277039